CLINICAL TRIAL: NCT03900442
Title: Phase 1 Pharmacodynamic and Pharmacokinetic Study of the Geranylgeranyltransferase I Inhibitor PTX-100 (GGTI-2418) in Patients With Advanced Malignancies
Brief Title: Phase 1 Study of PTX-100 in Patients With Advanced Malignancies With PTCL Expansion Cohort
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Prescient Therapeutics, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTX-100-PD-012017
Record Dates: First submitted 2019-03-13; First posted 2019-04-03 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Advanced Cancer; PTCL
Keywords: PTCL

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- PTX-100 (Experimental): IV infusion over 60 minutes on days 1 to 5 of a 14-day cycle for 4 cycles
  Interventions: Drug: PTX-100

INTERVENTIONS:
Drug: PTX-100 — Doses of 500 to 2000 mg/m2 will be administered.

SUMMARY:
This is an open-label, non-randomized study to evaluate the PD, PK, and safety of 500 to 2000 mg/m2 PTX-100 in patients with advanced malignancies.

PTX-100 will be administered by IV infusion over 60 minutes on days 1 to 5 of a 14-day cycle for 4 cycles unless toxicity is observed.

Dose escalation is complete and the expansion is open and actively recruiting PTCL patients.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy proven multiple myeloma (MM), peripheral T-cell lymphoma (CTCL, AITL or PTCL-NOS), colo-rectal cancer (CRC), pancreas cancer (PANC), or diffuse gastric cancer (DGC)
2. Must have a relapsed or refractory advanced malignancy for which no standard therapy exists.
3. Must have at least 6 unstained slides of archived formalin-fixed, paraffin-embedded tumor tissue available for genotyping studies; if insufficient or no archived tissue is available, a fresh tumor biopsy within 30 days prior to Cycle 1/Day 1 is mandatory.
4. Age ≥ 18 years
5. ECOG performance status ≤ 2
6. Adequate hematological function: absolute neutrophil count (ANC) ≥ 1000/mm3, platelet count ≥ 50,000 mm3
7. Adequate hepatic function: total bilirubin ≤ 1.5 times the upper limit of normal (ULN), and alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 times ULN (patients with liver metastases may be enrolled with elevated hepatic function based on Medical Monitor and Investigator review and agreement)
8. Adequate renal function: measured, calculated or estimated creatinine clearance of ≥ 50 mL/min
9. Female patients of childbearing potential must have a negative serum pregnancy test at screening and agree to use dual methods of contraception. Male patients must use an effective barrier method of contraception if sexually active with a female of childbearing potential. Acceptable methods of contraception are condoms with contraceptive foam, oral, implantable or injectable contraceptives, contraceptive patch, intrauterine device, diaphragm with spermicidal gel, or a sexual partner who is surgically sterilized or postmenopausal. For both male and female patients, effective methods of contraception must be used throughout the study and for 3 months following the last dose.
10. Informed consent (current IRB approved version) must be obtained from the patient or legally authorized representative prior to any study-related procedures.

Exclusion Criteria:

1. Radiation, chemotherapy, immunotherapy, or any other approved anticancer therapy ≤ 2 weeks prior to study treatment
2. Participation in another interventional investigational drug study within 4 weeks prior to enrollment
3. Concurrent radiation, chemotherapy, immunotherapy, or any other approved or investigational anticancer therapeutic (Patients are allowed to receive ≤ 10 mg/day corticosteroids for the treatment of non malignant disorders.)
4. Myocardial infarction within 6 months before screening, New York Heart Association Class II or greater heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, clinically significant pericardial disease, or electrocardiographic evidence of acute ischemic or active conduction system abnormalities
5. Uncontrolled infection requiring parenteral antibiotics, antivirals, or antifungals within 1 week prior to first dose (Patients with controlled infection or on prophylactic antibiotics are permitted in the study.)
6. Known to be HIV seropositive
7. Known active hepatitis A, B, or C infection or known to be positive for HCV RNA or HBsAg (HBV surface antigen)
8. Grade > 2 peripheral neuropathy at screening
9. Previous allogeneic transplant within the past 6 months or evidence of clinically significant graft-versus-host disease (if prior bone marrow transplant)
10. Any history of malignancy, other than that treated in this study, unless the patient has remained free of the disease for over 3 years (except for properly treated basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or breast)
11. Any active medical or psychiatric illness that, in the judgement of the investigator, may interfere with adherence to the protocol
12. Any malignancy with CNS involvement
13. History of allergic reactions attributed to compounds of similar chemical or biologic composition to PTX-100
14. Female patients who are pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-08-08 (Actual)

PRIMARY OUTCOMES:
Investigate the time- and dose-dependent PD of multiple doses of PTX-100 in patients with advanced malignancies (RAP-1) | One Cycle (cycle = 14 days)
  PD endpoints will be based on analysis of level of RAP-1 geranylgeranylation proteins in PBMNCs and tumor biopsies:
Investigate the time- and dose-dependent PD of multiple doses of PTX-100 in patients with advanced malignancies (PD endpoints) | One Cycle (cycle = 14 days)
  PD endpoints will be based on analysis of the level of DJ2 farnesylation proteins in PBMNCs and tumor biopsies:
Investigate the time- and dose-dependent PK of multiple doses of PTX-100 in patients with advanced malignancies (cmax) | One Cycle (cycle = 14 days)
  Pharmacokinetics will be evaluated by PK parameters calculated from plasma concentrations of PTX 100. Individual and mean plasma concentrations of PTX-100 versus time as well as individual and mean PK parameters will be determined, for the following:
  • Maximum observed plasma concentration (Cmax)
Investigate the time- and dose-dependent PK of multiple doses of PTX-100 in patients with advanced malignancies (Tmax) | One Cycle (cycle = 14 days)
  Pharmacokinetics will be evaluated by PK parameters calculated from plasma concentrations of PTX 100. Individual and mean plasma concentrations of PTX-100 versus time as well as individual and mean PK parameters will be determined, for the following:
  • Time to maximum observed plasma concentration (Tmax)
Investigate the time- and dose-dependent PK of multiple doses of PTX-100 in patients with advanced malignancies (half life) | One Cycle (cycle = 14 days)
  Pharmacokinetics will be evaluated by PK parameters calculated from plasma concentrations of PTX 100. Individual and mean plasma concentrations of PTX-100 versus time as well as individual and mean PK parameters will be determined, for the following:
  • Apparent elimination half-life (t1/2)

CONTACTS AND LOCATIONS:
Overall Officials: Terrence Chew, MD, Study Director — Prescient Therapeutics, Ltd.
Locations (1):
- Epworth Healthcare, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No